CLINICAL TRIAL: NCT00631436
Title: The Effects of Explosive Blast as Compared to Post-Traumatic Stress Disorder on Brain Function and Structure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center for Veterans Research and Education (Other)
Responsible Party: Scott Sponheim, Minneapolis VA Medical Center
Other Study IDs: PT074550; CDMRP PT074550
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2008-02

CONDITIONS: Blast Injuries; Traumatic Brain Injury; Post-Traumatic Stress Disorders
Keywords: Diffusion Tensor Imaging; Electroencephalography; Blast Injury; Traumatic Brain Injury
MeSH Terms: conditions — Blast Injuries; Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples and isolated DNA and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: If the individuals who meet the blast exposure criteria have a PCL score above 50 and meet the Hoge et al PCL criteria, thus indicating likely PTSD, they will be invited to participate as members of the Blast Exposed + PTSD group.
- 2: Other individuals meeting the blast exposure criteria will be invited to participate in the as members of the Blast Exposed + No PTSD group if they have PCL scores below 30.
- 3: Individuals reporting that they were not exposed to explosive blast will be recruited to participate. Those not exposed to blast but with PCL scores over 50 and meeting the Hoge et al PCL criteria will be invited to participate as members of the No Blast + PTSD group.
- 4: Individuals not exposed to blast with PCL scores below 30 will be invited to participate as members of the No Blast + No PTSD group.

SUMMARY:
Brain injury from explosive blast is a prominent feature of contemporary combat. Although protective armor and effective acute medical intervention allows soldiers to survive blast events, a growing number of veterans will have disability stemming from blast-related neural damage. Soldiers also return from combat with psychological disabilities caused by traumatic war events. The clinical presentation of individuals with blast-related neural damage and post-traumatic psychopathology are markedly similar and thus a clear description of the direct consequences of explosive blast is complicated by the emotional and cognitive sequelae of psychological trauma. We will use sophisticated measures of neural function and structure to characterize brain injury from explosive blasts in a sample of Operation Iraqi Freedom (OIF) National Guard soldiers who returned from deployment in the fall of 2007. Survey data gathered near the end of deployment indicated that over 50% of the brigade had been exposed to direct physical effects of explosive blasts. To fully characterize the effects of blast on the brain and differentiate them from post-traumatic stress disorder, we will contrast groups of soldiers exposed to blast and with groups experiencing post-traumatic stress disorder. This investigation will improve the characterization of blast-related traumatic brain injury, describe the essential features of the condition in terms of neural function and structure to inform diagnosis, and characterize mechanisms of recovery after blast-related neural injury to allow the creation of interventions that return soldiers to maximum levels of functioning.

DETAILED DESCRIPTION:
Background: The clinical presentation of individuals with blast-related brain injury and post-traumatic stress reactions can be markedly similar and thus a clear description of the direct consequences of explosive blast is complicated by the emotional and cognitive sequelae of psychological trauma. The inability to clearly separate the basis of symptoms for the two conditions has hampered clinicians in prescribing effective treatments that return soldiers to maximal functioning. Measures that directly assess neural disruption may be employed to differentiate blast-related brain injury from post-traumatic psychopathology and guide effective intervention..

Objective/Hypothesis: We propose to use quantitative indices of brain electrical activity and diffusion tensor imaging (DTI) to characterize the effects of blast injury on brain function and structure. We hypothesize that Operation Iraqi Freedom (OIF) soldiers injured by explosive blast will be distinguishable from those with post-traumatic stress disorder (PTSD) on measures of brain function and structure. Specifically, blast exposure will be associated with diminished P3a amplitudes to target stimuli during sustained attention and diminished lateralized frontal potentials during recognition of previously presented words. Individuals with PTSD will exhibit normal amplitudes of P3 and lateralized frontal brain potentials. Blast affected soldiers will also have compromised white matter integrity in supracallosal, inferior frontal, and superior frontal brain regions while PTSD will not be associated with these structural abnormalities. Finally, functional brain anomalies (e.g., P3a), and frontal white matter fractional anisotropy will be associated with the adaptive functioning of soldiers.

Specific Aims: Using advanced quantitative analyses of electroencephalogram recordings we will determine the nature of functional neural anomalies related to sustained attention and memory deficits evident after injury from blast. We will determine white matter anomalies that are unique to blast injury as compared to PTSD. We will also determine which aspects of blast-related functional and structural brain abnormalities are associated with adaptive functioning in post-deployment. The long-term goals for the proposed program of research are to improve the characterization of traumatic brain injury (TBI) due to blast, describe its essential features in terms of neural function and structure to improve diagnosis, and characterize mechanisms of recovery after blast-related neural injury to facilitate the creation of interventions that target pathophysiology.

Study Design: In May of 2007 over 2650 Minnesota National Guard troops of the 1/34 BCT completed a within-theatre survey on health, exposure to blast, and traumatic events. Fifty-one percent of surveyed troops reported being close enough to an explosive blast that they felt a heat or pressure wave, had trouble hearing, or had subsequent problems with attention or memory. The proposed study will be carried out over a four-year period and include a total of 180 subjects. To determine the neural consequences of blast exposure we will compare the functional and structural brain characteristics of individuals from the 1/34 BCT who have blast injury, blast injury and PTSD, PTSD, and no blast injury or PTSD. There will be 45 demographically similar subjects in each group.

ELIGIBILITY:
Inclusion Criteria:

* A high level of posttraumatic stress will be operationally defined "moderate" levels (a rating of 3 or more on a 1 to 5 scale) of the following symptoms according to Hoge et al 4: one re-experiencing symptom, three avoidance symptoms, and two hyperarousal symptoms. Staff will complete a screening interview via telephone in which the potential participant answers questions from the Blast Exposure Screen. The Blast Exposure Screen provides a comprehensive assessment of exposure to blast for the duration of deployment. Blast events will be rated for physical effects (e.g., knocked off balance, physically thrown by blast) and after effects (i.e., memory problems, headache) on the individual.
* Individuals who report memory lapses,
* Sensitivity to light or noise, headaches
* Difficulty with concentration shortly after the explosive blast and have any of the same symptoms in the past month will be invited to participate in the study.

Exclusion Criteria:

* Participants will be excluded from the study if they manifest
* Current substance induced psychotic disorder or psychotic disorder due to a general medical condition than TBI
* Current or past DSM IV defined substance dependence other than alcohol, caffeine, or nicotine
* Current DSM IV substance abuse other than alcohol, caffeine, or nicotine
* A neurologic condition or DSM Axis I mental disorder prior to deployment (predeployment data from a sample of soldiers from the 1/34 BCT yielded an estimated rate of 5% of either PTSD or depression)
* Current or predeployment unstable medical condition that would likely affect brain function (e.g., clear anoxic episode, cardiac arrest, current uncontrolled diabetes)
* Significant risk of suicidal or homicidal behavior
* Head injury from a source other than blast that resulted in loss of consciousness for more the 15 minutes, post-traumatic amnesia, skull fracture, or hospitalization. The screening interview will include questions to assess subjects with respect to the above exclusion criteria. During the telephone contact subjects will complete a screening for MRI protocols in order to exclude individuals who may have metal fragments in their bodies.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: National Guard Soldiers
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2008-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Sponheim, Ph.D., Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States